CLINICAL TRIAL: NCT05194553
Title: Identification and Characterization of Non-alcoholic Fatty Liver Disease Among Risk Groups in Turkey
Brief Title: Identification and Characterization of NAFLD in Turkey
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: Pax Clinic (Network)
Responsible Party: Sponsor
Other Study IDs: UMPAX-21-1
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver; Metabolic Syndrome; Overweight and Obesity
Keywords: NAFLD; fatty liver; NASH; non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver; Metabolic Syndrome; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is with 25% the most prevalent liver disorder in Western society and is associated with overweight, obesity, metabolic syndrome (MetS), type 2 diabetes mellitus (T2DM) and cardiovascular diseases (CVD). NAFLD is defined by a hepatic fat accumulation of more than 5% in the absence of classical causes of steatogenesis (e.g. alcohol and steatogenic drugs). It represents a broad spectrum of clinical entities from steatosis to advanced liver disease with hepatic failure. Most of the patients have simple steatosis, however in about 15-30% non-alcoholic steatohepatitis (NASH) develops, which leads to an overall increase in morbidity and mortality due to the progression to fibrosis, cirrhosis and hepatocellular carcinoma (HCC). Patients with NAFLD have no or few, mainly specific symptoms; and generally there is a silent progression of simple steatosis to NASH and in the end liver-related morbidity and mortality. Despite the clinical importance and the potential impact on healthcare resources, the majority of NAFLD patients are currently not detected due to the lack of non-invasive methods to diagnose NAFLD. To date, the prevalance of NAFLD in Turkey among subjects at risk, and its relation to common comorbidities such as obesity, T2DM and CVD is not clear. Therefore, identification of NAFLD patients in this cohort will give information on the prevalence in the group of uncomplicated overweight and obesity and those with concomitant cardiometabolic diseases. By early detecting these patients at risk to develop progressive liver diseases and extrahepatic manifestations, it will be possible to intervene and improve health. Within this context, this study aims to detect prevalence of NAFLD among risk groups. Also, the risk factors related to NAFLD etiology and progression, such as overweight, obesity, T2DM, CVD, diet and physical activity will be studied to have a better understanding of their presumed causal relationship with NAFLD.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD), characterized with more than 5% intrahepatic fat accumulation in the absence of classical causes of steatogenesis, is considered as a growing epidemic with a global prevalence estimated around 25%. NAFLD usually manifests as simple steatosis, however in about 15-30% cases it can progress to its inflammatory type of NASH, which may in turn lead to fibrosis, cirrhosis, and hepatocellular carcinoma (HCC). Given that patients typically have no or few symptoms, it is fundamental to detect and treat NAFLD at the earliest stage to decrease liver-related morbidity and mortality.

NAFLD is known to be the hepatic manifestation of the metabolic syndrome (MetS), a cluster of metabolic disorders including abdominal obesity, type 2 diabetes mellitus (T2DM), and cardiovascular diseases (CVD). It has been reported that NAFLD risk increases with obesity, diabetes mellitus, and dyslipidemia. In line with this, the highest prevalence of NAFLD is reported from South America and the Middle East, where MetS is also widespread, making it a major public health issue in these regions. Similarly, the clinical significance of NAFLD has progressively increased in Turkey lately. With an obesity rate of 32% according to latest WHO reports, and T2DM rate of 15%, Turkey can be considered a risky region in terms of NAFLD burden. Despite the increasing burden of NAFLD in Turkey, few studies have been undertaken to identify its prevalence showing conflicting results due to excessive heterogeneity in design. 8 studies that were undertaken in the past 15 years reported a prevalence between 10,6% and 60%. One study that included subjects with MetS reported as high as 94.3%. It is critically important to develop new evidence regarding NAFLD prevalence among this patient group in Turkey and the association between MetS comorbidities and NAFLD severity so as to establish NAFLD risk groups and develop effective population screening and public health policies targeting this patient group.

The optimal screening method to detect hepatic steatosis in the general population remains to be established. The reference standard is liver biopsy; however, it is problematic to conduct studies that involve liver biopsy due to its invasiveness, high cost and patient discomfort. Therefore, ultrasonographic imaging (USG) is usually favored as the first-line modality in most clinical practices. However, USG has limited sensitivity and does not reliably detect steatosis when <20% or in individuals with BMI>40 kg/m2. Controlled attenuation parameter (CAP) measured with transient elastography (TE), on the other hands, has recently emerged as a reliable imaging tool for the screening and diagnosis of NAFLD on a population scale. It is suggested to have high sensitivity in identifying mild steatosis and yields a good correlation with steatosis grades. Therefore, CAP can enable early and noninvasive detection of NAFLD at the subclinical level. It is important to detect NAFLD at the earliest possible stage because once it is established hepatic insulin resistance increases, which, in turn, may trigger, in 30-40% of cases, NAFLD progression to its inflammatory phenotype Non-alcoholic Steatohepatitis (NASH) and eventually, hepatocarcinoma, cirrhosis, and liver failure.

As of today, treatment of NAFLD is only possible through lifestyle modifications such as following a healthy balanced diet and doing regular physical activity, given that no pharmacological treatment has been approved yet for NAFLD. Weight loss of 7-10% BW seems to have proven efficacy especially in overweight subjects. Different dietetic approaches have been proposed to reach the weight loss goal; however, no consensus has been reached yet on the type of medical nutrition therapy to be offered to NAFLD patients. Having said that, in the recent EASL-EASD-EASO Clinical Practice Guidelines, Mediterranean diet (MED DIET) was recommended as the diet of choice for the treatment of NAFLD together with weight loss initiatives. Indeed, a growing body of evidence suggest that MED DIET exerts health benefits even without accompanying weight reduction, which is the main obstacle in lifestyle interventions.

Higher adherence to the MED DIET has shown to have beneficial effects on the progression of hepatic steatosis in observational studies and clinical trials (n<90 followed up for<6 months) in patients with existing hepatic steatosis. These findings are confirmed in The Swiss CoLaus and UK Fenland cohorts which reported lower risk of hepatic steatosis with higher adherence to MED DIET.

Not only the dietary pattern, but also certain micronutrient deficiencies might be related to NAFLD. New evidence suggests that also Vitamin D deficiency, which is known to associate with obesity and sedentary lifestyle, may cause NAFLD. Hypovitaminosis D is proposed to have a causative relationship with the severity and incidence of NAFLD. The association between Hypovitaminosis D and NAFLD has been examined previously. A lower serum 25(OH)D level was shown to be an independent risk factor for NAFLD. Various studies has shown a correlation between Vitamin D level and disease severity. A cross-sectional study of 6567 men concluded that participants in the lowest tertile of serum 25(OH)D levels had a significantly increased risk for NAFLD compared to those in the highest tertile. Another study found similar results. CAP was used as a tool to define hepatic steatosis in a study that showed a significant association between serum 25(OH)D levels and NAFLD.9 However, some other studies reported quite contradictory results. Collectively, the data from the published studies indicate that NAFLD subjects are more likely to be vitamin D deficient compared to controls. However, definite directionality of the results cannot be ascertained due to the limitations which include the variability in the method of diagnosis of NAFLD, clinical heterogeneity among the study groups and variability in defining vitamin D deficiency. Demonstration of a causal role of hypovitaminosis D in NAFLD progress could have important therapeutic implications. Vitamin D supplementation is easy to accomplish on a population level, hence, it can be an efficient tool to prevent NAFLD. Cochrane performed a systematic review of randomized clinical trials of Vitamin D supplementation in chronic liver diseases, 11 of which included NAFLD patients. Given the high heterogeneity of studies included, they failed to assess the beneficial and harmful effects of vitamin D supplementation in adults with chronic liver diseases. Well-designed future studies are needed to investigate this potential relation.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign the informed consent
* Able to speak Turkish
* Between 18-80 years
* BMI >25 kg/m²
* Having one of the following conditions: 1)Insulin resistance 2)Impaired glucose tolerence 3)type 2 diabetes mellitus, 4)hypertension 5)dyslipidemia 6)cardiovascular diseases (atherosclerosis, angina pectoris, ischaemic heart condition, cerebrovascular condition)

Exclusion Criteria:

* Excessive alcohol use (more than 20 g/day for women and 30g/day for men= >2 glasses alcohol/day for women and >3 glasses for men)
* Other liver diseases: Hepatitis B virus, Hepatitis C virus, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, Wilson's disease, Alpha 1 antitrypsin deficiency
* Secondary causes for steatosis: disorders of lipid metabolism, HCV Genotype 3, total parental nutrition, severe surgical weight loss, medications (amiodarone, tamoxifen, methotrexate, corticosteroids and HAART), lean steatosis, Celiac disease, environmental toxicity
* Pregnancy and breastfeeding.
* A history of bariatric surgery.
* Diagnosis of liver cirrhosis and/or hepatocellular carcinoma.
* Current diagnosis of extrahepatic malignancy(s) or prior diagnosis within last 5 years.
* Individuals about to undergo a surgery or otherwise medical procedure that will interfere with data collection and analyses planned within the current cohort, will initially be excluded from participation, but are offered the opportunity to participate at a later moment in time (e.g., after 3 months are myocardial infarction patients are eligible for participation).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 500 male and female participants aged between 18-80, who can sign the informed consent and are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
prevalence of NAFLD in risk groups in Turkey | 1 year

SECONDARY OUTCOMES:
NAFLD's relation to risk factor: overweight | 1 year
  To see if there is an effect of having a BMI between 25 and 30 kg/m² in the development of NAFLD. The physiological parameter used will be BMI.
NAFLD's relation to risk factor: obesity | 1 year
  To see if there is an effect of having a BMI more than 30 kg/m² in the development of NAFLD. The physiological parameter used will be BMI.
NAFLD's relation to risk factor: IR | 1 year
  To see if there is an effect of having a HOMA-IR more than 2.5 in the development of NAFLD. The physiological parameter used will be HOMA-IR.
NAFLD's relation to risk factor: T2DM | 1 year
  Type 2 diabetes mellitus will be assessed based on previous diagnosis and HbA1c levels.
NAFLD's relation to risk factor: HT | 1 year
  To see if there is an effect of Hypertension in the development of NAFLD. The physiological parameter used will be systolic and diastolic blood pressure.
NAFLD's relation to risk factor: MetS | 1 year
  To see if there is an effect of metabolic syndrome (defined by the criteria of the International Diabetes Federation) on the development of NAFLD.
NAFLD's relation to risk factor: CVD | 1 year
  Cardiovascular diseases will be assessed based on medical history found in the patient files.
NAFLD's relation to risk factor: PAL | 1 year
  Physical Activity Level will be determined based in IPAQ mini results
NAFLD's relation to VDD | 1 year
  To see if there is an effect of Vitamin D deficiency in the development of NAFLD. The physiological parameter used will be 25(OH)Vit D.
NAFLD's relation to Med Diet adherence | 1 year
  To see if there is an effect of Mediterranean Diet adherence in the development of NAFLD. The parameter used will be Med Diet adherence screening scale (MEDAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Pax Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided